CLINICAL TRIAL: NCT02050672
Title: Effect of Myoinositol Treatment of Spermatozoa on in Vitro Fertilization Outcome: a Prospective, Randomized Sibling-oocyte Study
Brief Title: Effect of Myoinositol Treatment of Spermatozoa on in Vitro Fertilization Outcome
Acronym: MI_ICSI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AGUNCO Obstetrics and Gynecology Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: MI_ICSI
Record Dates: First submitted 2014-01-27; First posted 2014-01-31 (Estimated); Last update posted 2021-08-06 (Actual); Status verified 2021-07

CONDITIONS: Couple Sterility
Keywords: Myoinositol; ART; EMBRYO QUALITY
MeSH Terms: interventions — Inositol

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- untreated (Active Comparator): Semen was prepared with routinely used media
  Interventions: Other: untreated
- myo-inositol (Experimental): routinely used semen preparation media have been enriched with myo-inositol 2mg/ml.
  in particular the stock solution was prepared in order to add 15microliters per ml of medium
  Interventions: Dietary Supplement: Myo-inositol

INTERVENTIONS:
Dietary Supplement: Myo-inositol
  Arms: myo-inositol
Other: untreated
  Arms: untreated

SUMMARY:
In the present trial, the investigators aim to evaluate whether semen myo-inositol (MI) treatment is able to improve IVF outcomes.

In particular, retrieved oocytes will be randomly divided in two groups, one group will be inseminated with MI treated semen while the other will be inseminated with untreated semen.

DETAILED DESCRIPTION:
Myo is synthesized from glucose-6-phosphate, it is a precursor of second messengers in the cell signaling pathways and it is involved in the regulation of intracellular calcium.

Literature data have demonstrated the MI play a crucial role in reproduction, indeed, oocyte and spematozoa are nursed in a medium congaing hig MI concentration.

Furthermore, it has been demonstrated that, in oligoasthenoteratozoospermic patients, in vitro incubation with 2 mg/ml of myo increase significantly the number of spermatozoa with high mitochondrial membrane potential (MMP). Moreover, it has been found that the in vitro fertilization rate is correlated with the percentage of high MMP spermatozoa.

ELIGIBILITY:
Inclusion Criteria:

* couple counselled for IVF

Exclusion Criteria:

* cryopreserved sample

Ages: 30 Years to 42 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 249 (Actual)
Dates: Start 2013-05; Primary Completion 2021-01 (Actual); Study Completion 2021-07 (Actual)

PRIMARY OUTCOMES:
Fetilization rate | Day 1

SECONDARY OUTCOMES:
Embryo quality | Day 2 to Day 5

CONTACTS AND LOCATIONS:
Locations (1):
- TECNOLAB, Milan, Italy

REFERENCES:
- [Background] Condorelli RA, La Vignera S, Bellanca S, Vicari E, Calogero AE. Myoinositol: does it improve sperm mitochondrial function and sperm motility? Urology. 2012 Jun;79(6):1290-5. doi: 10.1016/j.urology.2012.03.005. PMID 22656408
- [Background] Nomikos M, Swann K, Lai FA. Starting a new life: sperm PLC-zeta mobilizes the Ca2+ signal that induces egg activation and embryo development: an essential phospholipase C with implications for male infertility. Bioessays. 2012 Feb;34(2):126-34. doi: 10.1002/bies.201100127. Epub 2011 Nov 16. PMID 22086556
- [Background] Condorelli RA, La Vignera S, Di Bari F, Unfer V, Calogero AE. Effects of myoinositol on sperm mitochondrial function in-vitro. Eur Rev Med Pharmacol Sci. 2011 Feb;15(2):129-34. PMID 21434479